CLINICAL TRIAL: NCT04864834
Title: A 52-week Multicenter, Randomized, Double-masked, 2-arm Parallel Study to Compare Efficacy, Safety and Immunogenicity of SOK583A1 to Eylea®, Administered Intravitreally, in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Phase III Study Assessing the Efficacy, Safety and Immunogenicity of SOK583A1 Versus Eylea® in Patients With Neovascular Age-related Macular Degeneration
Acronym: Mylight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSOK583A12301
Record Dates: First submitted 2021-04-15; First posted 2021-04-29 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-07

CONDITIONS: Neovascular Age-related Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOK583A1 (40 mg/mL) (Experimental): Intravitreal (IVT) administration of 2 mg of SOK583A1 in the study eye, every 4 weeks (q4w) at Baseline, Week 4 and Week 8, and thereafter every 8 weeks (q8w) at week 16, 24, 32, 40 and 48.
  Interventions: Biological: SOK583A1 (40 mg/mL)
- Eylea EU (40 mg/mL) (Active Comparator): IVT administration of 2 mg of Eylea EU in the study eye, every 4 weeks (q4w) at Baseline, Week 4 and Week 8, and thereafter every 8 weeks (q8w) at week 16, 24, 32, 40 and 48.
  EU: European
  Interventions: Biological: Eylea EU (40 mg/mL)

INTERVENTIONS:
Biological: SOK583A1 (40 mg/mL) — IVT administration of 2 mg of SOK583A1 in the study eye, every 4 weeks (q4w) at Baseline, Week 4 and Week 8, and thereafter every 8 weeks (q8w) at week 16, 24, 32, 40 and 48.
  Arms: SOK583A1 (40 mg/mL)
Biological: Eylea EU (40 mg/mL) — IVT administration of 2 mg of Eylea EU in the study eye, every 4 weeks (q4w) at Baseline, Week 4 and Week 8, and thereafter every 8 weeks (q8w) at week 16, 24, 32, 40 and 48.
  Arms: Eylea EU (40 mg/mL)

SUMMARY:
Purpose and rationale: To demonstrate similar efficacy, safety and immunogenicity of SOK583A1 and Eylea EU as per Eylea approved treatment regimen in patients with nAMD.

The primary clinical question of interest is: Does SOK583A1 have similar efficacy as Eylea EU in terms of mean change in BCVA score in participants with nAMD who are anti-VEGF naive, without important protocol deviations and adherent to the treatment and completed the treatment to Week 8?

DETAILED DESCRIPTION:
BCVA: Best-Corrected Visual Acuity Eylea EU: Europe-authorized Eylea® nAMD: Neovascular Age-related Macular Degeneration VEGF: Vascular Endothelium Growth Factor

ELIGIBILITY:
Participants eligible for inclusion in this study must meet all of the following criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Participants must be 50 years of age or older at Screening
3. Anti-VEGF treatment-naive patients for either eye and systemically
4. Study eye diagnosed with active CNV lesions (type 1 and/ or type 2) secondary to AMD and/or Retinal Angiomatous Proliferation lesions (type 3), affecting the central subfield. Active CNV lesion is defined by the presence of leakage as evidenced by fluorescein angiography, and intra- or subretinal fluid as evidenced by optical coherence tomography, both confirmed by the CRC at Screening
5. Total area of CNV (including both classic and occult components) must comprise > 50% of the total lesion area in the study eye, confirmed by the CRC at Screening
6. BCVA between 73 and 38 letters, both inclusive, in the study eye at Screening and Baseline using ETDRS testing charts
7. Willing and able to comply with all study procedures, and be likely to complete the study
8. Clear ocular media and adequate pupil dilatation in both eyes to permit good quality photographic imaging.

Participants meeting any of the following criteria are not eligible for inclusion in this study.

Ocular conditions and treatments:

1. Previous treatment with any anti-VEGF therapy in either eye or investigational drugs in study eye or fellow eye, at any time prior to Baseline
2. Participant has received any approved treatment for nAMD (other than vitamin and dietary supplements) in the study eye and at any time prior to Baseline
3. Presence of other causes of CNV, including pathologic myopia (spherical equivalent of -8 diopters or more negative), ocular histoplasmosis syndrome, angioid streaks,choroidal rupture, or multifocal choroiditis in the study eye, assessed by imaging at screening by CRC and appropriately stated in the multi-modal eligibility confirmation report
4. Any active or suspected intraocular or periocular infection or suspected active intraocular inflammation (e.g infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in either eye at Screening or Baseline
5. Subfoveal fibrosis, atrophy, or scarring extending > 50% of total lesion area in the study eye as assessed by the Investigator at Screening and confirmed by the CRC prior to randomization
6. Subretinal hemorrhage that is ≥ 50% of the total lesion area in the study eye, or if the subretinal hemorrhage involving the fovea is 1 or more disc areas (≥ 2.54 mm2 ) in size in the study eye, as assessed by Fluorescein Angiography (FA) and confirmed by the CRC
7. Retinal pigment epithelium (RPE) rip/tear in the study eye at Screening or Baseline
8. Current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Baseline
9. History or evidence of the following, in the study eye:

   * Intraocular (including cataract surgery) or refractive surgery within the 90 day period prior to Baseline. The yttrium aluminum garnet (YAG) posterior capsulotomy is allowed no later than 4 weeks prior to Baseline
   * Previous penetrating keratoplasty or vitrectomy
   * Previous panretinal photocoagulation
   * Previous photodynamic therapy
   * Previous submacular surgery or other surgical intervention for AMD
   * Retinal detachment or treatment or surgery for retinal detachment
   * Any history of macular hole of stage 2 and above
   * Prior trabeculectomy or other filtration surgery
   * Ocular trauma within the 6-months period prior to Baseline
10. History of hypersensitivity to any of the study treatments or its excipients, or clinically relevant sensitivity to fluorescein dye, as assessed by the Investigators
11. Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication or according to Investigator's judgment at Screening or Baseline
12. Aphakia and/or absence of the posterior capsule in the study eye at Screening or Baseline, unless it occurred as a result of a YAG posterior capsulotomy in association with prior posterior chamber intraocular lens implantation
13. Intra or periocular use of corticosteroids in the study eye within a 6 month period prior to Baseline
14. Use of topical ocular corticosteroids in the study eye for 30 or more consecutive days within the 90 days period prior to Baseline
15. Previous therapeutic radiation near the region of the study eye
16. Concomitant conditions or ocular disorders in the study eye, including media opacities, cataract and diabetic macular edema, at Screening or Baseline which could, in the opinion of the Investigator, prevent response to study treatment or may confound interpretation of study results (efficacy and safety), compromise visual acuity or require medical or surgical intervention during the course of the study
17. Presence of amblyopia, amaurosis or ocular disorders with BCVA <38 letters (ETDRS testing charts) in the fellow eye at Screening (except when due to conditions whose surgery may improve VA, e.g. cataract)
18. Presence of Scleromalacia in either eye
19. Participants requiring anti-VEGF treatment of the fellow eye at Baseline will not be eligible for the PK substudy

    Systemic conditions and treatments:
20. Previous systemic treatment with any anti-VEGF therapy
21. Use of systemic corticosteroids for 30 or more consecutive days within the 90 days prior to Baseline, with the exception of low stable doses of corticosteroids (defined as ≤ 10 mg prednisolone or equivalent dose used for 90 days or more).
22. Uncontrolled blood pressure defined as a systolic value ≥ 160 mmHg or diastolic value ≥ 100 mmHg at Screening
23. Stroke or myocardial infarction during the 6-month period prior to Baseline
24. Participation in an investigational systemic drug, biologic, or device study within 30 days or duration of 5 half-lives of the investigational product (whichever is longer) prior to Baseline. Note: observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary
25. Presence of infection at screening or active infection within 2 weeks before screening
26. Underlying advanced, severe and uncontrolled concomitant condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, inflammatory, infectious or gastrointestinal), physical examination finding, or clinical laboratory finding which in the opinion of the Investigator place the participant at unacceptable risk from participation in the study
27. History of a medical condition (including, but not limited to chronic disease immunosuppression, metabolic dysfunction, prior exposure to other drugs that may pose risk of infection or allergic reactions) that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product, or that might affect participant safety or interpretation of the study results.
28. Pregnant or nursing (lactating) women and women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 3 months after stopping the medication. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.
    * Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2023-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (28):
  - Sandoz Investigational Site, Phoenix, Arizona
  - Sandoz Investigational Site, Arcadia, California
  - Sandoz Investigational Site, Campbell, California
  - Sandoz Investigational Site, Encino, California
  - Sandoz Investigational Site, Fullerton, California
  - Sandoz Investigational Site, Glendale, California
  - Sandoz Investigational Site, Huntington Beach, California
  - Sandoz Investigational Site, Pasadena, California
  - Sandoz Investigational Site, Poway, California
  - Sandoz Investigational Site, Redlands, California
  - Sandoz Investigational Site, Sacramento, California
  - Sandoz Investigational Site, Fort Myers, Florida
  - Sandoz Investigational Site, Pinellas Park, Florida
  - Sandoz Investigational Site, Plantation, Florida
  - Sandoz Investigational Site, Stuart, Florida
  - Sandoz Investigational Site, Marietta, Georgia
  - Sandoz Investigational Site, Oak Forest, Illinois
  - Sandoz Investigational Site, Hagerstown, Maryland
  - Sandoz Investigational Site, Albuquerque, New Mexico
  - Sandoz Investigational Site, Great Neck, New York
  - Sandoz Investigational Site, Liverpool, New York
  - Sandoz Investigational Site, Rochester, New York
  - Sandoz Investigational Site, Eugene, Oregon
  - Sandoz Investigational Site, Rapid City, South Dakota
  - Sandoz Investigational Site, Abilene, Texas
  - Sandoz Investigational Site, Arlington, Texas
  - Sandoz Investigational Site, Willow Park, Texas
  - Sandoz Investigational Site, Lynchburg, Virginia
- Australia (6):
  - Sandoz Investigational Site, Albury, New South Wales
  - Sandoz Investigational Site, Liverpool, New South Wales
  - Sandoz Investigational Site, Parramatta, New South Wales
  - Sandoz Investigational Site, Sydney, New South Wales
  - Sandoz Investigational Site, Adelaide, South Australia
  - Sandoz Investigational Site, Melbourne, Victoria
- Austria (2):
  - Sandoz Investigational Site, Linz, Upper Austria
  - Sandoz Investigational Site, Graz
- Sandoz Investigational Site, Sofia, Bulgaria
- Czechia (2):
  - Sandoz Investigational Site, Pardubice
  - Sandoz Investigational Site, Prague
- France (3):
  - Sandoz Investigational Site, Marseille, Bouches-Du-Rhone
  - Sandoz Investigational Site, Saint-Cyr-sur-Loire, Indre Et Loire
  - Sandoz Investigational Site, Paris
- Germany (7):
  - Sandoz Investigational Site, Düsseldorf
  - Sandoz Investigational Site, Frankfurt am Main
  - Sandoz Investigational Site, Freiburg im Breisgau
  - Sandoz Investigational Site, Hanover
  - Sandoz Investigational Site, Leipzig
  - Sandoz Investigational Site, Mainz
  - Sandoz Investigational Site, Marburg
- Hungary (7):
  - Sandoz Investigational Site, Budapest, HUN
  - Sandoz Investigational Site, Budapest, Pest County
  - Sandoz Investigational Site, Budapest
  - Sandoz Investigational Site, Debrecen
  - Sandoz Investigational Site, Sopron
  - Sandoz Investigational Site, Szeged
  - Sandoz Investigational Site, Székesfehérvár
- Israel (7):
  - Sandoz Investigational Site, Haifa
  - Sandoz Investigational Site, Jerusalem
  - Sandoz Investigational Site, Kfar Saba
  - Sandoz Investigational Site, Lod
  - Sandoz Investigational Site, Petah Tikva
  - Sandoz Investigational Site, Rehovot
  - Sandoz Investigational Site, Tel Aviv
- Japan (12):
  - Sandoz Investigational Site, Nagakute, Aichi-ken
  - Sandoz Investigational Site, Nagoya, Aichi-ken
  - Sandoz Investigational Site, Fukuoka, Fukuoka
  - Sandoz Investigational Site, Kure, Hiroshima
  - Sandoz Investigational Site, Amagasaki, Hyōgo
  - Sandoz Investigational Site, Kobe, Hyōgo
  - Sandoz Investigational Site, Inashiki-gun, Ibaraki
  - Sandoz Investigational Site, Kagoshima, Kagoshima-ken
  - Sandoz Investigational Site, Hamamatsu, Shizuoka
  - Sandoz Investigational Site, Meguro-ku, Tokyo
  - Sandoz Investigational Site, Taito-ku, Tokyo
  - Sandoz Investigational Site, Ube, Yamaguchi
- Sandoz Investigational Site, Riga, Latvia
- Lithuania (2):
  - Sandoz Investigational Site, Kaunas, Kaunas County
  - Sandoz Investigational Site, Vilnius
- Poland (5):
  - Sandoz Investigational Site, Krakow, Malopolska
  - Sandoz Investigational Site, Bydgoszcz
  - Sandoz Investigational Site, Lodz
  - Sandoz Investigational Site, Lublin
  - Sandoz Investigational Site, Wroclaw
- Portugal (2):
  - Sandoz Investigational Site, Coimbra
  - Sandoz Investigational Site, Porto
- Slovakia (3):
  - Sandoz Investigational Site, Žilina, Slovak Republic
  - Sandoz Investigational Site, Bratislava
  - Sandoz Investigational Site, Trenčín
- Spain (6):
  - Sandoz Investigational Site, Bilbao, Basque Country
  - Sandoz Investigational Site, Sant Cugat del Vallès, Catalonia
  - Sandoz Investigational Site, Pamplona, Navarre
  - Sandoz Investigational Site, Oviedo, Principality of Asturias
  - Sandoz Investigational Site, Barcelona
  - Sandoz Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 485 subjects were randomized in the study, and 484 subjects received at least 1 dose of SOK583 or Eylea EU and comprised the Safety Set. Of these 484 subject, 1 subject in the SOK583 group had no post-baseline BCVA assessments and was therefore excluded from the Full Analysis Set. The Full Analysis Set therefore comprises 483 subjects.
Groups:
- Eylea EU (40 mg/mL): IVT administration of 2 mg of Eylea EU in the study eye, every 4 weeks (q4w) at Baseline, Week 4 and Week 8, and thereafter every 8 weeks (q8w) at week 16, 24, 32, 40 and 48.
  EU: European
  Eylea EU (40 mg/mL): IVT administration of 2 mg of Eylea EU in the study eye, every 4 weeks (q4w) at Baseline, Week 4 and Week 8, and thereafter every 8 weeks (q8w) at week 16, 24, 32, 40 and 48.
Period: Overall Study
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Started | 245 | 240
Safety Set | 244 | 240
Full Analysis Set | 243 | 240
Per-Protocol Set | 235 | 226
PK Analysis Set | 23 | 20
Immunogenicity Analysis Set | 234 | 231
VEGF Analysis Set | 60 | 67
Completed | 216 | 215
Not Completed | 29 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL) | Total
Number analyzed (Participants) | 243 | 240 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.8 (7.82) | 75.7 (7.72) | 75.7 (7.76)
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 103 | 98 | 201
  ≥75 years | 140 | 142 | 282
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 136 | 273
  Male | 106 | 104 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 9 | 21
  Not Hispanic or Latino | 225 | 225 | 450
  Unknown or Not Reported | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 12 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 215 | 214 | 429
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 42 | 88
  Europe | 158 | 161 | 319
  Australia | 10 | 13 | 23
  Israel | 15 | 12 | 27
  Japan | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Best-Corrected Visual Acuity (BCVA) Will be Assessed Using the ETDRS Testing Charts at an Initial Distance of 4 Meters. The Change From Baseline in BCVA in Letters is Defined as Difference Between BCVA Score Between Week 8 and Baseline.
Description: The primary aim of the study is to demonstrate equivalence of change in BCVA score from Baseline at Week 8 between participants with nAMD treated with SOK583A1 and participants treated with Eylea EU. The primary analysis will be performed on the Per-Protocol Set (PPS), which is the most appropriate analysis set to use when testing for equivalence.
  ETDRS: Early Treatment Diabetic Retinopathy Study EU: European
Time Frame: Change from baseline in mean BCVA score at Week 8
Population: Per-Protocol Set
Measure: Mean (Standard Deviation); unit: BCVA score in letters
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 235 | 226
BCVA score in letters | 6.5 (8.98) | 6.8 (7.46)

2. Secondary Outcome: Similarity in the Anatomical Outcome Between SOK583A1 and Eylea EU
Description: Mean change in CSFT using SD-OCT from Baseline to Week 1, 4, 8, 24 and 52
  CSFT: Central Subfield Thickness SD-OCT: Spectral-Domain Optical Coherence Tomography
Time Frame: Week 1, 4, 8, 24 and 52
Population: Full Analysis Set (subjects with baseline value). Results are provided for subjects with data available at a certain visit.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 243 | 238
μm
  Week 1: number analyzed (Participants) | 227 | 229
  Week 1 | -103.6 (89.91) | -99.2 (86.18)
  Week 4: number analyzed (Participants) | 240 | 231
  Week 4 | -152.9 (123.55) | -140.7 (120.25)
  Week 8: number analyzed (Participants) | 240 | 232
  Week 8 | -165.7 (144.35) | -154.2 (133.43)
  Week 24: number analyzed (Participants) | 233 | 227
  Week 24 | -136.4 (140.19) | -127.5 (137.87)
  Week 52: number analyzed (Participants) | 224 | 224
  Week 52 | -187.9 (150.70) | -172.9 (142.74)

3. Secondary Outcome: Similarity in the Anatomical Outcome Between SOK583A1 and Eylea EU
Description: Mean change of CNV lesion size using FA from Screening to Week 8 and 52
  CNV: Choroidal neovascularization FA: Fundus Angiography
Time Frame: Week 8 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 242 | 237
mm^2
  Week 8: number analyzed (Participants) | 223 | 218
  Week 8 | -1.7877 (3.97567) | -1.7274 (3.77398)
  Week 52: number analyzed (Participants) | 205 | 211
  Week 52 | -3.7845 (5.21911) | -3.5026 (4.96036)

4. Secondary Outcome: Similarity of Efficacy Between SOK583A1 and Eylea EU in Terms of BCVA
Description: Mean change from Baseline in BCVA score using EDTRS testing charts at Week 24 and 52
Time Frame: Week 24 and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 243 | 240
score on a scale
  Week 24: number analyzed (Participants) | 234 | 229
  Week 24 | 6.9 (8.93) | 7.4 (9.95)
  Week 52: number analyzed (Participants) | 227 | 227
  Week 52 | 6.4 (11.91) | 7.7 (11.62)

5. Secondary Outcome: Similarity Between SOK583A1 and Eylea EU in Terms of Safety
Description: Number and proportion of subjects with ocular and non-ocular Adverse Events (AEs) over 52 weeks including serious AEs, regardless of relationship to study treatment
Time Frame: 52 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 244 | 240
Participants
  Ocular AEs in the study eye | 84 | 78
  Ocular AEs in the fellow eye | 55 | 51
  Non-ocular AEs | 141 | 141

6. Secondary Outcome: Similarity Between SOK583A1 and Eylea EU in Terms of Immunogenicity
Description: Development of binding and neutralizing Anti-drug antibodies (ADAs) up to Week 52
Time Frame: Week 52
Population: Immunogenicity analysis set including all randomized subjects who received at least 1 dose of study treatment and had immunogenicity blood samples collected and analyzed at baseline and at least 1 post-baseline time point. Subjects with positive ADA results at baseline were excluded from the IAS. Subjects who received both treatments into the study eye were excluded from the IAS. Subjects were analyzed according to the study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 234 | 231
Participants
  ADA positive | 2 | 6
  ADA negative | 232 | 225

7. Secondary Outcome: Systemic Exposure to SOK583A1 and Eylea EU in Participants of the Pharmacokinetic (PK) Assessment
Description: Aflibercept concentration assessments at Baseline (pre-dose) and 24 hours after the first and third injections
Time Frame: Baseline (pre-dose) and 24 hours after the first injection (day 2) and third injection (day 58)
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 23 | 20
ng/ml
  Day 1 (Baseline): number analyzed (Participants) | 21 | 20
  Day 1 (Baseline) | 0.0 (0.0) | 0.0 (0.0)
  Day 2: number analyzed (Participants) | 21 | 20
  Day 2 | 32.0 (24.0) | 33.3 (24.6)
  Day 58: number analyzed (Participants) | 22 | 17
  Day 58 | 31.7 (21.9) | 33.6 (25.8)

8. Other Pre Specified Outcome: Analysis Systemic VEGF Concentrations in Patients Treated With Aflibercept
Description: Mean VEGF concentrations
Time Frame: Assessment at Week 48 (pre-dose) and Week 52
Population: VEGF Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | SOK583A1 (40 mg/mL) | Eylea EU (40 mg/mL)
Number analyzed (Participants) | 60 | 67
pg/mL
  Week 48 (pre-dose): number analyzed (Participants) | 57 | 62
  Week 48 (pre-dose) | 86.44 (77.962) | 80.09 (92.155)
  Week 52 | 75.14 (20.892) | 73.38 (20.169)

ADVERSE EVENTS:
Time Frame: 52 weeks
Groups:
- SOK583: SOK583
- Eylea EU: Eylea EU
Arm/Group | SOK583 | Eylea EU
All-Cause Mortality (participants affected / at risk) | 5/244 | 1/240
Serious Adverse Events (participants affected / at risk) | 39/244 | 30/240
Other Adverse Events (participants affected / at risk) | 58/244 | 63/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOK583 (N=244) | Eylea EU (N=240)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 2 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vitreoretinal traction syndrome (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 3 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOK583 (N=244) | Eylea EU (N=240)
Neovascular age-related macular degeneration (Eye disorders) | 25 | 25
Visual acuity reduced (Eye disorders) | 11 | 12
COVID-19 (Infections and infestations) | 19 | 23
Hypertension (Vascular disorders) | 11 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Sandoz agreements with its investigators may vary. However, Sandoz does not prohibit any investigators from publishing. Any publications from a single-site are postponed until the publication of the pooled date (i.e. data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04864834/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04864834/SAP_001.pdf